CLINICAL TRIAL: NCT02854605
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability, and Efficacy of GS-9674 in Subjects With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Evaluating the Safety, Tolerability, and Efficacy of GS-9674 in Participants With Nonalcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-402-1852; 2016-002496-10 (EudraCT Number)
Record Dates: First submitted 2016-07-29; First posted 2016-08-03 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
Keywords: Non-alcoholic fatty liver disease (NAFLD); Fibrosis; GS-9674
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GS-9674 30 mg (Experimental): GS-9674 30 mg + placebo to match GS-9674 100 mg for 24 weeks
  Interventions: Drug: GS-9674; Drug: Placebo to match GS-9674
- GS-9674 100 mg (Experimental): GS-9674 100 mg + placebo to match GS-9674 30 mg for 24 weeks
  Interventions: Drug: GS-9674; Drug: Placebo to match GS-9674
- Placebo (Placebo Comparator): Placebo to match GS-9674 30 mg + placebo to match GS-9674 100 mg for 24 weeks
  Interventions: Drug: Placebo to match GS-9674

INTERVENTIONS:
Drug: GS-9674 — Tablet administered orally once daily
  Arms: GS-9674 100 mg; GS-9674 30 mg
Drug: Placebo to match GS-9674 — Tablet(s) administered orally once daily

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of GS-9674 in participants with nonalcoholic steatohepatitis (NASH).

ELIGIBILITY:
Key Inclusion Criteria:

* Meets the following conditions:

  * A clinical diagnosis of nonalcoholic fatty liver disease (NAFLD)
  * Screening magnetic resonance imaging - proton density fat fraction (MRI-PDFF) with ≥ 8% steatosis
  * Screening magnetic resonance elastography (MRE) with liver stiffness ≥ 2.5 kilopascal (kPa) OR
  * A historical liver biopsy within 12 months of screening consistent with NASH with fibrosis, but not cirrhosis, and
  * No documented weight loss > 5% between the date of the liver biopsy and screening.
* Platelet count ≥ 150,000/mm^3
* Albumin ≥ 3.3 g/dL
* Serum creatinine ≤ upper limit of normal (ULN)

Key Exclusion Criteria:

* Pregnant or lactating females
* Alanine aminotransferase (ALT) > 5x upper limit of the normal range (ULN)
* Other causes of liver disease including autoimmune, viral, and alcoholic liver disease
* Cirrhosis of the liver

  * Prior history of decompensated liver disease, including ascites, hepatic encephalopathy, or variceal bleeding
* Body mass index (BMI) < 18 kg/m^2
* Uncontrolled diabetes mellitus (hemoglobin A1c > 9% at screening)
* International normalized ratio (INR) > 1.2 unless on anticoagulant therapy
* Total bilirubin > 1 x ULN, except with diagnosis of Gilbert's syndrome

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (37):
- United States (26):
  - Ruane Clinical Research Group Inc., Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Inland Empire Liver Foundation, Rialto, California
  - Clinical Research of South Florida, Coral Gables, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Northwestern Memorial Hospital, Clinical Research Unit, Chicago, Illinois
  - Crescent Clinical Research Center, LLC, Metairie, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Kansas City Research Institute, Kansas City, Missouri
  - Concorde Medical Group, PLLC, New York, New York
  - Duke University Medical Center, Duke South Clinics, Durham, North Carolina
  - Carolinas Center for Liver Disease/Carolinas HealthCare System, Durham, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Gastro One, Germantown, Tennessee
  - Quality Medical Research, PC, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Texas Digestive Disease Consultants, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Pinnacle Clinical Research, Live Oak, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - Intermountain Liver Disease and Transplant Center, Murray, Utah
  - Bon Secours St. Mary's Hospital of Richmond, Inc d/b/a Bon Secours Liver Institute of Virginia, Newport News, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Inc. d/b/a Bon Secours Liver Institute of Virginia, Richmond, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Swedish Organ Transplant and Liver Center, Seattle, Washington
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - LMC Clinical Research Inc (Bayview), Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Liver Center, Toronto, Ontario
  - Toronto Digestive Disease Associates, Inc., Vaughan, Ontario
- Hong Kong (2):
  - Princess Margaret Hospital, Kowloon
  - The Chinese University of Hong Kong, Shatin
- Auckland Clinical Studies, Auckland, New Zealand
- Switzerland (2):
  - Universitatsspital Bern, Inselspital, Universitatsklinik fur Viszerale Chirurgie und Medizin, Hepatologie, Bern
  - Universitatsspital Zurich, Zurich
- Addenbrooke's Hospital, Cambridge, United Kingdom

REFERENCES:
- [Derived] Patel K, Harrison SA, Elkhashab M, Trotter JF, Herring R, Rojter SE, Kayali Z, Wong VW, Greenbloom S, Jayakumar S, Shiffman ML, Freilich B, Lawitz EJ, Gane EJ, Harting E, Xu J, Billin AN, Chung C, Djedjos CS, Subramanian GM, Myers RP, Middleton MS, Rinella M, Noureddin M. Cilofexor, a Nonsteroidal FXR Agonist, in Patients With Noncirrhotic NASH: A Phase 2 Randomized Controlled Trial. Hepatology. 2020 Jul;72(1):58-71. doi: 10.1002/hep.31205. PMID 32115759

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Hong Kong, New Zealand, and Europe. The first participant was screened on 26 October 2016. The last study visit occurred on 09 January 2018.
Pre-assignment Details: 327 participants were screened.
Groups:
- GS-9674 100 mg: GS-9674 100 mg tablet once daily + placebo-to-match (PTM) GS-9674 30 mg tablet once daily for 24 weeks.
- GS-9674 30 mg: GS-9674 30 mg tablet once daily + PTM GS-9674 100 mg tablet once daily for 24 weeks.
- Placebo: PTM GS-9674 30 mg tablet once daily + PTM GS-9674 100 mg tablet once daily for 24 weeks.
Period: Overall Study
Arm/Group | GS-9674 100 mg | GS-9674 30 mg | Placebo
Started | 56 | 56 | 28
Completed | 53 | 49 | 24
Not Completed | 3 | 7 | 4
Not completed — Adverse Event | 1 | 5 | 2
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Withdrew Consent | 1 | 0 | 1
Not completed — Investigator's Discretion | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- GS-9674 100 mg: GS-9674 100 mg tablet once daily + PTM GS-9674 30 mg tablet once daily for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | GS-9674 100 mg | GS-9674 30 mg | Placebo | Total
Number analyzed (Participants) | 56 | 56 | 28 | 140
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55 (10.5) | 51 (12.8) | 50 (9.9) | 53 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 15 | 87
  Male | 21 | 19 | 13 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 19 | 8 | 44
  Not Hispanic or Latino | 39 | 37 | 20 | 96
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, Customized: American Indian or Alaska Native | 0 | 1 | 1 | 2
  Race, Customized: Asian | 13 | 5 | 4 | 22
  Race, Customized: Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Race, Customized: Black or African American | 1 | 1 | 1 | 3
  Race, Customized: White | 42 | 47 | 21 | 110
  Race, Customized: Other | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 1 | 2 | 1 | 4
  Canada | 12 | 7 | 6 | 25
  Hong Kong | 5 | 2 | 3 | 10
  United States | 37 | 43 | 16 | 96
  United Kingdom | 1 | 0 | 0 | 1
  Switzerland | 0 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Safety of GS-9674 as Assessed By Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as 1 or both of the following: 1) Any adverse events (AE) with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug, 2) Any AEs leading to premature discontinuation of study drug.
Time Frame: Up to 24 weeks plus 30 days
Population: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | GS-9674 100 mg | GS-9674 30 mg | Placebo
Number analyzed (Participants) | 56 | 56 | 28
Percentage of participants
  TEAEs | 89.3 | 76.8 | 67.9
  TEAEs leading to premature discontinuation of drug | 1.8 | 8.9 | 7.1

2. Primary Outcome: Overall Safety of GS-9674 as Assessed By Percentage of Participants With Treatment-Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any post-baseline time point, up to and including the date of last dose of study drug plus 30 days for participants who permanently discontinued study.
Time Frame: Up to 24 weeks plus 30 days
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | GS-9674 100 mg | GS-9674 30 mg | Placebo
Number analyzed (Participants) | 56 | 56 | 28
Percentage of participants
  Any Grade ≥ 1 | 89.3 | 92.9 | 92.9
  Grade 1 | 35.7 | 42.9 | 50.0
  Grade 2 | 37.5 | 37.5 | 25.0
  Grade 3 | 7.1 | 10.7 | 14.3
  Grade 4 | 8.9 | 1.8 | 3.6

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Arm/Group | GS-9674 100 mg | GS-9674 30 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56 | 0/28
Serious Adverse Events (participants affected / at risk) | 2/56 | 2/56 | 1/28
Other Adverse Events (participants affected / at risk) | 39/56 | 34/56 | 17/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GS-9674 100 mg (N=56) | GS-9674 30 mg (N=56) | Placebo (N=28)
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GS-9674 100 mg (N=56) | GS-9674 30 mg (N=56) | Placebo (N=28)
Vertigo (Ear and labyrinth disorders) | 3 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 5 | 1
Constipation (Gastrointestinal disorders) | 1 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 4 | 2
Fatigue (General disorders) | 2 | 7 | 1
Bronchitis (Infections and infestations) | 3 | 3 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3 | 3
Sinusitis (Infections and infestations) | 1 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 5 | 2
Urinary tract infection (Infections and infestations) | 4 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 2
Headache (Nervous system disorders) | 4 | 6 | 4
Depression (Psychiatric disorders) | 1 | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 9 | 5
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 | 3 | 0
Hypertension (Vascular disorders) | 3 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (4):
  • Study Protocol: Original (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT02854605/Prot_000.pdf
  • Study Protocol: Amendment 1 (2016-10-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT02854605/Prot_001.pdf
  • Study Protocol: Amendment 2 (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT02854605/Prot_002.pdf
  • Statistical Analysis Plan (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT02854605/SAP_003.pdf